CLINICAL TRIAL: NCT05633641
Title: Clinical Study of Peripheral Blood Neoantigen Specific T Cells Predicting the Efficacy of Immunotherapy for Esophageal Squamous Cell Carcinoma
Brief Title: Peripheral Blood Neoantigen Specific T Cells Predict the Efficacy of Immunotherapy for Esophageal Squamous Cell Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xianghua Wu, Principal Investigator, Fudan University
Other Study IDs: TAS-T- 20220328
Record Dates: First submitted 2022-11-21; First posted 2022-12-01 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a single-center clinical and exploratory study. Peripheral blood tumor antigen-specific T lymphocytes of patients with resectable esophageal cancer treated with neoadjuvant chemotherapy combined with immunotherapy and patients with advanced or metastatic esophageal cancer treated with first-line chemotherapy were detected at different time points to predict ORR after neoadjuvant chemotherapy combined with immunotherapy for resectable esophageal cancer and pCR rate, DFS after radical resection and first-line metastasis of advanced esophageal cancer Therapy combined with immunotherapy for ORR, PFS and OS.

ELIGIBILITY:
Inclusion Criteria:

.Volunteer to participate in clinical studies and sign informed consent. .Aged 18-70 years, expected survival > 3 months. .Gender: Male or female. .Locally advanced esophageal squamous cell carcinoma and metastatic esophageal .squamous cell carcinoma.

.There should be at least one measurable lesion (diameter ≥10 mm according to RECIST standards, and those that have undergone TACE or ablative treatment and met the requirements by imaging can be used as the target lesion).

.ECOG Physical state score 0-1.

* Laboratory test results within one week before enrollment meet the following conditions:
* White blood cells (WBC) ≥ 3.0x10 ^9 /L.
* Neutrophils (ANC) ≥ 1.5x10 ^9 /L (without G-CSF support).
* Platelets ≥100 x10^9/L.
* Hemoglobin ≥100 g/L (no blood transfusion support within 7 days).
* Prothrombin time ≤1.5x upper limit time (about 14 seconds).
* Serum creatinine <2.5 mg/dl or < 1.5 times the normal high value for that age.
* Endogenous creatinine clearance ≥50 ml/min.
* Serum total bilirubin ≤ 1.5x normal high value.
* Serum alkaline phosphatase ≤ 2.5x normal high value.
* Serum aspartate aminotransferase (AST) ≤2.5x normal high value.
* Serum glutalanine aminotransferase (ALT) ≤2.5x normal high value.
* Lactate dehydrogenase level (LDH) determination.
* Determination of serum immunoglobulin content.
* Determination of serum β2 microglobulin level.
* Serum virus (CMV, EBV, HBV, HCV) negative.

Exclusion Criteria:

.Diseases of vital organs (e.g., cardiovascular and respiratory systems) : myocardial infarction, myocardial ischemia, history of coronary artery bypass or symptoms of coronary ischemia, obstructive or restrictive lung disease.

.The patient has poor immune tolerance and may be less responsive to immune cell therapy or prone to toxic reactions.

.Previous autoimmune and immune deficiency diseases. .Radiotherapy pneumonia. .Oxygen dependent individuals. .Other therapeutic studies or clinical trials were enrolled within four weeks. The experimental vaccine was administered within two months. .Systemic use of glucocorticoids, hydroxyurea or immunosuppressants (such as IL-2, IFN-α, IFN-γ, GSF, mTOR inhibitors, cyclosporine, etc.) within two weeks. Except for those who have recently or are currently using inhaled hormones.

.Chronic or recurrent severe autoimmune disease within one year. .There is an uncontrolled active infection. .2-4 during acute or persistent graft-versus-host disease (GVHD). .Patients with severe heart disease, whose condition remained unstable after treatment, had myocardial infarction, congestive heart failure, unstable angina pectoris, pericardial effusion with obvious symptoms or unstable arrhythmia within 6 months before enrollment.

.Coagulopathy. .HIV infection.

* Previous history of other cancers excluding:
* Patients with basal cell carcinoma or squamous cell carcinoma with active treatment and complete wound healing.
* Cure of cervical or breast carcinoma in situ for at least three years.
* The primary malignancy was completely resected and in complete remission for 5 years or more.

.Brain metastases with symptoms of cranial hypertension. Remarks: Patients with brain metastases who have been effectively treated are eligible for admission.

.Persons with Intellectual Disabilities. .Suspected or confirmed history of alcohol and drug abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: locally advanced esophageal squamous cell carcinoma and advanced esophageal squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-10-19 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ORR | until 1 year or recurrence
  objective response rate

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer hospital Fudan University, Shanghai, Shanghai Municipality, China